CLINICAL TRIAL: NCT07226596
Title: Advancing Non-Abstinence Outcomes in the Treatment of Methamphetamine Use Disorder
Brief Title: Non-Abstinence Outcomes in Methamphetamine Use Disorder
Acronym: RCT (05)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 107171; R01DA064144 (NIH)
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Methamphetamine Use Disorder
Keywords: methamphetamine; treatment; behavioral intervention

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will receive payment for providing urine samples throughout the trial.
- Contingency Management Group (Experimental): This group will receive payment for providing methamphetamine negative urine samples throughout the trial.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Subjects will receive payments for providing methamphetamine negative urine samples.
  Arms: Contingency Management Group

SUMMARY:
Reduced drug use is a clinically meaningful target for treatment development, but few studies have evaluated the positive impacts produced by this behavioral change, preventing adoption of this endpoint in clinical trials. The proposed research will fill that critical knowledge gap by demonstrating the biopsychosocial benefits of reduced methamphetamine use. These data will be used to change current accepted methamphetamine treatment endpoints and accelerate identification of therapies for methamphetamine use disorder.

ELIGIBILITY:
Inclusion Criteria:

* be age 18 years or older;
* self-report methamphetamine use in the week prior to screening;
* provide a methamphetamine-positive urine sample at screening;
* meet DSM-5 criteria for moderate-severe Methamphetamine Use Disorder (MUD);
* be seeking treatment for their methamphetamine use
* be able and willing to commit to the 12-week intervention, as well as the 12-week post-intervention follow-up
* Individuals who meet these criteria and are stably maintained on buprenorphine or methadone for Opioid Use Disorder (OUD) will also be eligible to participate.

Exclusion Criteria:

* current or past medical or psychiatric illness (e.g., physical dependence on any drug other than buprenorphine requiring medically managed detoxification, unstable angina, uncontrolled cardiac arrhythmia, aortic stenosis, self-reported compromised immune function, severe diagnosis for a SUD other than MUD or treated OUD) that would interfere with study participation in the opinion of the study physicians
* poor venous access precluding blood draws

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2031-01-04 (Estimated); Study Completion 2031-01-04 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Pressure | At baseline.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 1 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 2 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 3 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 4 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 5 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 6 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 7 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 8 of participation.
  Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 8 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 9 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 10 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 11 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Mean Arterial Pressure | Week 12 of participation.
  Mean Arterial Pressure is recorded during subject visits and is recorded in mm Hg
Endothelin-1 | At baseline.
  Endothelin-1 levels will be measured. They will be recorded in pg/ml.
Endothelin-1 | Week 6 of participation.
  Endothelin-1 levels will be measured. They will be recorded in pg/ml.
Endothelin-1 | Week 12 of participation.
  Endothelin-1 levels will be measured. They will be recorded in pg/ml.

SECONDARY OUTCOMES:
Sleep | At baseline.
  Sleep will be measured with the Pittsburgh Sleep Quality Index, with a range from 0-21 where lower scores are better.
Sleep | Week 4 of participation.
  Sleep will be measured with the Pittsburgh Sleep Quality Index, with a range from 0-21 where lower scores are better.
Sleep | Week 8 of participation.
  Sleep will be measured with the Pittsburgh Sleep Quality Index, with a range from 0-21 where lower scores are better.
Sleep | Week 12 of participation.
  Sleep will be measured with the Pittsburgh Sleep Quality Index, with a range from 0-21 where lower scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Psychopharmacology of Addiction Laboratory, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant level data will be findable and identifiable using the unique number assigned to this grant application by NIDA. Where the data are available and how to access the data will be identified in any publications and presentations about these data. The repository and funding source will also be acknowledged in any publications and presentations. The Open Science Framework, which is a generalist repository, will be the data repository. This repository has policies and procedures in place that will provide data access to qualified researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: No later than one year after the completion of the funded project period. Data will be available indefinitely after that.
Access Criteria: Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and could be used for secondary study purposes.